CLINICAL TRIAL: NCT06900972
Title: Effect of Colloids Versus Crystalloids on Heart Mechanics: a Double-blind Cross Over Randomized Trial
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Nidhal Bouchahda, Dr Nidhal Bouchahda, University of Monastir
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TN2025-NAT-INS-125
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Fluid Reponsiveness; Fluid Resuscitation; Fluid Therapy
Keywords: colloids; cristalloids; heart mechanics
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AB (Other): Patients will blindly receive colloids then after a washout period of 7 days a cristalloids solute will be administered
  Interventions: Drug: Gelafundin; Drug: Saline (NaCl 0,9 %) (placebo)
- BA (Other): Patients will blindly receive cristalloids then after a washout period of 7 days a colloids solute will be administered.
  Interventions: Drug: Gelafundin; Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: Gelafundin — Volunteers will undergo a comprehensive transthoracic echocardiography to measure left ventricular torsion, global longitudinal strain, left atrial strain and free wall right ventricular strain before any intervention. Initially, 500 ml of the specified but blinded solution will be administered, followed by a repeat of the echocardiographic process. Subsequently, an additional 500 ml will be given, totaling 1000 ml, and strain curves will be reacquired. After a washout period of 7 days, the same procedure will be repeated with the second solution.
Drug: Saline (NaCl 0,9 %) (placebo) — Volunteers will undergo a comprehensive transthoracic echocardiography to measure left ventricular torsion, global longitudinal strain, left atrial strain and free wall right ventricular strain before any intervention. Initially, 500 ml of the specified but blinded solution will be administered, followed by a repeat of the echocardiographic process. Subsequently, an additional 500 ml will be given, totaling 1000 ml, and strain curves will be reacquired. After a washout period of 7 days, the same procedure will be repeated with the second solution

SUMMARY:
The debate over whether to use colloid or crystalloid solutions for fluid resuscitationis still ongoing. Colloid solutions consist of large molecules that generally cannot pass through healthy capillary membranes, whereas crystalloid solutions contain ions that easily move from the intravascular space to the interstitial compartment. Therefore, it is traditionally argued that colloids are more effective at expanding intravascular volume, with a suggested ratio of 1:3 compared to crystalloids. However, there is currently limited evidence to suggest that resuscitation with one type of fluid is more effective or safer than t he other. Despite these theoretically advantageousphysiological properties, colloids have not demonstrated a clear hemodynamic benefit over crystalloids. We hypothesized that these unexpected discrepancies may be attributed to different mechanical heart responses.

ELIGIBILITY:
Inclusion Criteria:

* HealthyVolunteers with age > 18 years without medical history

Exclusion Criteria:

History of cardio vascular diseases Diabetes Hypertension Currentpregnancy Knownallergy to one of the tested products Leftventricular dysfunction discovered at baseline assessment Valvular heart or other structural diseases discovered at base line assessment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Heart mechanics response will be assessed by using left ventricular longitudinal strain, left ventricular torsion strain curves, left atrial strain curves and right ventricular free wall strain curves | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Fattouma Bourguiba Hospital, Monastir, Tunisia, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Myburgh JA, Mythen MG. Resuscitation fluids. N Engl J Med. 2013 Sep 26;369(13):1243-51. doi: 10.1056/NEJMra1208627. No abstract available. PMID 24066745